CLINICAL TRIAL: NCT01924715
Title: Evaluating the Cost Effectiveness of ISTDP: A Quasi Experimental Study
Acronym: CEISTDP
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: AA003
Record Dates: First submitted 2013-07-25; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-07

CONDITIONS: Anxiety; Somatoform Disorders; Personality Disorders; Depression; Psychotic Disorders
Keywords: somatoform disorder; psychotherapy; depression; anxiety; personality disorder
MeSH Terms: conditions — Anxiety Disorders; Somatoform Disorders; Personality Disorders; Depression; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ISTDP: Patients provided Intensive Short term Dynamic Psychotherapy
  Interventions: Behavioral: ISTDP
- Control Group: Patients referred for ISTDP but never seen for any reason

INTERVENTIONS:
Behavioral: ISTDP — An emotion focused brief psychotherapy format.
  Other Names: Intensive Short-term Dynamic Psychotherapy
  Groups: ISTDP

SUMMARY:
Objective: To evaluate whether or not cases treated with Intensive Short-term Dynamic Psychotherapy (ISTDP) facilitate healthcare cost reduction, whether any observed reduction is greater than that of a control group and whether any such gains would be maintained in follow up.

Design: A quasi-experimental design was employed in which pre and post healthcare cost and usage data were extracted for all ISTDP treated cases from 1999 to 2008 and compared to parallel measures of a control group of cases referred but never treated.

DETAILED DESCRIPTION:
Importance: Psychiatric and psychological disorders result in excess health care service use and costs. Brief psychotherapy methods may be effective across a broad range of mental disorders and could therefore result in healthcare cost reduction.

Objective: To evaluate whether or not cases treated with Intensive Short-term Dynamic Psychotherapy (ISTDP) facilitate healthcare cost reduction, whether any observed reduction is greater than that of a control group and whether any such gains would be maintained in follow up.

Design: A quasi-experimental design was employed in which pre and post healthcare cost and usage data were extracted for all ISTDP treated cases from 1999 to 2008 and compared to parallel measures of a control group of cases referred but never treated.

Setting: Treatments were provided at an urban University based psychotherapy service.

Participants: All cases from the province of Nova Scotia treated within the research time frame were included. 890 patients were included with a very broad range of psychiatric disorders including anxiety, mood, somatoform, personality and psychotic disorders. 192 referred but never see cases served as non randomized controls.

Intervention(s): ISTDP is an emotionally focused form of brief psychotherapy which has supportive, cognitive, experiential and primarily psychodynamic elements. In this setting the average length of treatment was 7.3 sessions and cost an estimated $500 dollars per treatment course.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for ISTDP treatment

Exclusion Criteria:

* Patients not referred for ISTDP treatment

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Major DSM IV categories included including mood, anxiety, personality, somatoform, dissociative, eating and psychotic disorders
Sampling Method: Non-Probability Sample
Enrollment: 1082 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Total Doctor and Hospital Costs | 1 year pre versus 3 years post
  Total Physician and Hospital billings per patient

SECONDARY OUTCOMES:
Hospital costs | 1 year pre versus 3 years post
  Total Hospital costs per patient
Hospital Days | 1 year per versus 3 years post
  Hospital days per patient
Doctor Visits | 1 year pre versus 3 years post
  Doctor Costs per patient
Doctor Costs | 1 year pre versus 3 years post
  Doctor costs per patient

CONTACTS AND LOCATIONS:
Overall Officials: Allan A Abbass, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Abbass A, Kisely S, Rasic D, Town JM, Johansson R. Long-term healthcare cost reduction with Intensive Short-term Dynamic Psychotherapy in a tertiary psychiatric service. J Psychiatr Res. 2015 May;64:114-20. doi: 10.1016/j.jpsychires.2015.03.001. Epub 2015 Mar 25. PMID 25840829